CLINICAL TRIAL: NCT05347810
Title: Comfort During Prolonged Exposure to Repetitive Forces Mimicking Exoskeleton Use
Brief Title: Comfort Thresholds for Repetitive Forces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roessingh Research and Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 80800
Record Dates: First submitted 2022-03-29; First posted 2022-04-26 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Exoskeleton; Safety; Comfort; physical Human-Robot Interaction

STUDY DESIGN:
Intervention Model Description: The study is a cross-sectional intervention study with one measurement session, where participants will provide a continuous comfort rating during exposure to repetitive normal and shear forces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All participants in the study will receive the same investigational treatment (application of prolonged repetitive forces) and provide continuous comfort ratings.
  Interventions: Other: Application of repetitive forces mimicking exoskeleton use

INTERVENTIONS:
Other: Application of repetitive forces mimicking exoskeleton use — The investigational treatment consists of applying a predefined set of continuous and repetitive forces to the participant's thigh. It is applied using a custom device that has been designed specifically for this study. The forces to be applied are based on forces measured during exoskeleton use and will not exceed pain pressure thresholds reported in literature. The participants will hold an enabling switch at all times which they can activate to release the force exerted to their thigh. Alternatively, the experimenter can activate an emergency switch if the situation seems unsafe.

SUMMARY:
Exoskeletons can be used for rehabilitation, as assistive device for patients, or to support workers during strenuous tasks. To fulfil their purpose, they need to apply forces to the user's musculoskeletal system. The forces are transmitted at skin level through an interface, often in the form of cuffs. Adverse events causing discomfort and injuries to the skin and underlying tissue can be attributed to those interaction forces. While there is some information about safe limit values for impact forces or pressure and shear applied for short durations, little is known regarding comfort and safety thresholds for repetitive forces applied over long durations as is the case in exoskeleton use. This study therefore aims at gaining new knowledge on safe and limit values, based on discomfort (staying below pain threshold), for continuous repetitive shear and normal forces applied through a cuff.

Therefore, the primary objective is to determine comfort thresholds for prolonged exposure to repetitive normal and shear stress exerted to the human thigh via a cuff with straps, using different force patterns comparable to those exerted during exoskeleton use. The secondary objectives are to determine the feasibility of the experiment, the influence of subject characteristics on comfort thresholds, the occurrence of skin injuries or other negative signs, and whether characteristics of muscle activity can be related to discomfort.

DETAILED DESCRIPTION:
Rationale: Exoskeletons can be used for rehabilitation, as assistive device for patients, or to support workers during strenuous tasks. To fulfil their purpose, they need to apply forces to the user's musculoskeletal system. The forces are transmitted at skin level through an interface, often in the form of cuffs. Adverse events causing discomfort and injuries to the skin and underlying tissue can be attributed to those interaction forces. While there is some information about safe limit values for impact forces or pressure and shear applied for short durations, little is known regarding comfort and safety thresholds for repetitive forces applied over long durations as is the case in exoskeleton use. This study therefore aims at gaining new knowledge on safe and limit values, based on discomfort (staying below pain threshold), for continuous repetitive shear and normal forces applied through a cuff.

Objective: The primary objective is to determine comfort thresholds for prolonged exposure to repetitive normal and shear stress exerted to the human thigh via a cuff with straps, using different force patterns comparable to those exerted during exoskeleton use. The secondary objectives are to determine the feasibility of the experiment, the influence of subject characteristics on comfort thresholds, the occurrence of skin injuries or other negative signs, and whether characteristics of muscle activity can be related to discomfort.

Study design: The study is a cross-sectional intervention study with one measurement session, where participants will provide a continuous comfort rating during exposure to repetitive normal and shear forces.

Study population: The aim is to include 20 healthy participants in total, matching the age groups 18-35 and 55-85.

Intervention: A pre-defined set of prolonged repetitive force patterns will be applied to each participant's thigh though a contact force which is similar to cuffs commonly used in gait exoskeletons. The forces will be applied by a custom made actuated test device and are based on normal use of exoskeletons.

Main study parameters/endpoints: The main study parameter is the level of discomfort as indicated continuously by the participants through a slider with a visual analogue scale. The scale reaches from no discomfort at all to maximum imaginable discomfort. A separate switch which releases all forces if activated by the participant is used to detect onset of pain.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study is non-therapeutic, so no direct benefits for the participants are involved. The procedures are non-invasive and safety measures are taken to avoid excessive force exertion to the participants or other unsafe situations. Therefore, subjects suffer no negative effects or disadvantages, except for the invested time and the discomfort experienced during the force execution. Pain will be avoided as participants can trigger a release of the forces at any time. Any changes to the participants' skin or other negative signs will be monitored and followed up on until they have resolved.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 35 or between 55 and 85 years of age
* Able to provide informed consent

Exclusion Criteria:

* Unable to follow simple instructions
* Insufficient knowledge of the Dutch or English language to understand the purpose and methods of the study
* skin lesions at the thigh
* sensory impairments
* severe blood pressure fluctuations
* inability to sit in required posture in experiment chair for 60 minutes
* taking blood thinners or showing signs for increased bleeding tendency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Perceived discomfort as indicated on a 10 mm visual analog scale (VAS) by the participants, ranking from 'no discomfort' to 'worst imaginable comfort' (10) | 80 minutes
  The level of discomfort will be indicated on a VAS as a percentage of maximum imaginable discomfort through a slider that is positioned within reach of the subjects. It will be synchronized with the forces exerted in relation to time. The onset of discomfort, i.e. the point at which the slider of the VAS is first moved to a position >0, is recorded as discomfort detection threshold (DDT). If the participant activates the enabling switch indicating that the force creates pain rather than discomfort, this point is recorded as pain detection threshold (PDT).

SECONDARY OUTCOMES:
Number of completed test sessions/dropouts | 160 minutes
  To investigate feasibility and tolerability of experiments
Occurrence of injuries or other negative signs | 30 minutes
  Records of skin changes directly after the sessions and short structured interview on the phone 2-4 days after the intervention
Surface Electromyography (EMG) recordings of Rectus femoris | 120 minutes
  Muscle activity

OTHER OUTCOMES:
Height in meters | 2 minutes
  Height and weight will later be combined to report BMI in kg/m²
Body weight in kg | 2 minutes
  Height and weight will later be combined to report BMI in kg/m²
Age in years | 1 minute
  Age will reported as one subject characteristic
Gender | 1 minute
  Gender will be reported as one subject characteristic

CONTACTS AND LOCATIONS:
Overall Officials: Gerdienke Prange, PhD, Principal Investigator — Roessingh Research and Development
Locations (1):
- Roessingh Research and Development, Enschede, Netherlands

IPD SHARING:
Plan to Share IPD: No